CLINICAL TRIAL: NCT05011591
Title: Effects of Manipulating Swimming Speed and Frequency on Swimming Economy in High-level Swimmers and Para-swimmers
Brief Title: Swimming Economy in Swimmers and Paraswimmers as a Function of SR(Stroke Rate) and V(Velocity) Manipulations (NePTUNE-3)
Acronym: NePTUNE-3
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Rouen Normandie (Other)
Collaborators: French Institute of Sport (INSEP) (Unknown); French swimming federation (FFN) (Unknown); French federation of handisport (Unknown)
Responsible Party: Principal Investigator, Letocart Adrien, Project manager, University of Rouen Normandie
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: URouenNormandie
Record Dates: First submitted 2021-07-22; First posted 2021-08-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Swimming; Coordination Lack; Oxygen Consumption; Lactic Acid Blood Increased
Keywords: swimming economy; Para-swimmers; Athletes; Energetics; coordination
MeSH Terms: conditions — Ataxia; Hyperlactatemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- swimming economy (Experimental): This is a study based on a comparative clinical trial (effect of an imposed V and/or SR on the swimming economy of swimmers or para-swimmers). This longitudinal study is carried out on a representative sample of swimmers and para-swimmers selected for their potential at the Paris 2024 Olympic and Paralympian Games. Following a standardized warm-up, all swimmers will perform intermittent swimming tests of progressive velocity in a 50 m indoor pool in their swimming specialty with or without an imposition of the SR to adopt. During the trials, the swimmers and para-swimmers will be equipped with inertial measurement units, as well as a heart rate monitor and tissue oximeters. The swimming and non-swimming phases will also be filmed continuously. Gas exchanges will be recorded 2 minutes after the warm-up and during the 7 minutes of passive recovery. Micro blood samples will be taken from the earlobe at the end of the warm-up and at 1, 3, 5 and 7 minutes of recovery between each trial.
  Interventions: Other: Swimming economy

INTERVENTIONS:
Other: Swimming economy — Detailed in arm's section

SUMMARY:
The competitive swimming and open water swimming events are scheduled for the 2024 Paris Olympic and Paralympian Games. Generally associated with a non-neglectable number of medals in the last Olympics, swimming performance depends on the swimmer's ability to manage his or her Stroke Length and Stroke Rate, where Velocity can be defined as the product of SR and SL. The optimisation of this management depends on the swimmer's ability to develop a large motor repertoire and to use the coordination mode (catch-up, opposition, superposition) best suited to the environmental constraints and opponents' adversity. These adaptations may contribute to 1) a modification of the energy expenditure or be dependent on the energy supply necessary for muscular contraction and 2) the preferential use of one or other of the metabolic pathways in the production of this chemical energy, moreover in an aquatic environment inducing particular thermal exchanges.

DETAILED DESCRIPTION:
To swim fast, one need to be able to create great propelling forces in addition to minimizing resistance. Propulsion emerged from the appropriate spatial-temporal coordination of the four limbs. The purpose of this study is to determine the motor repertoire (coordination possibilities) of each swimmer and para-swimmer in order to monitor their swimming economy, as a function of their energy expenditure. Crawl coordination has been studied extensively, and recent technologies such as inertial units and machine learning methods may be combined to characterize it automatically. There is a strong need to extend this knowledge to the other three swimming strokes and adapt it to para-swimmers' disabilities to clearly measure the impacts of SR and V manipulations on swimming economy.

Swimming is performed in a complex aquatic environment serving both as a support for propulsion and as a resistance to progress forward. Therefore, to properly behave through water, swimmers coordinate their limbs to increase their velocity (V). Cyclic activities performance, such as swimming, corresponds to the reaching of high speed, defined by the product of stroke length (SL, in m.cycle-1) and stroke frequency (SR, cycles.min-1). Many authors have therefore focused on the behaviors of elite swimmers and they observed a change in arm coordination when values of 1.8 m.s-1 in V and/or 50 cycles.min-1 in SR were reached. Such results are related to the high degree of flexibility in the swimmer's motor behavior , that should not imply an additional energy expenditure that may become detrimental to performance. Studies showed that changes in V and/or SR would influence the value of the energy cost of swimming. These studies, mainly performed in front crawl would be of valuable interest to develop for all other strokes (i.e. breaststroke, butterfly and backstroke) and for multiple group of participants (i.e. para-swimmers).

Two intermittent swimming tests of progressive velocity will be performed in the swimmers' and para-swimmers' specialty with or without prescription of the SR. Coordination and physiological variables will be collected to investigate if changes in motor behaviors are linked to changes in energy expenditure.

The study will be performed in two main centers, with a duration of the inclusion period equals to 3 years. Moreover, the duration of participation of each participant is also fixed to 3 years . One of the objectives is obtaining a landscape of possible motor behaviors for each participant according to the manipulation of swimming frequency and speed. This 'landscape' will show whether, for all participants, the behavioral adaptations are efficient (in reference to their energy expenditure).

ELIGIBILITY:
Inclusion Criteria:

* High-level swimmers and para-swimmers on ministerial lists
* Current license to participate in national and international competitions
* Over 12 and under 50 years old
* Signed consent form
* Willingness to participate / cooperate

Exclusion Criteria:

* Absence of authorization from legal guardians for the minor athlete at the time of inclusion in the study.
* For disabled athletes: non-union fracture, pressure sore stage 2 or more, infection (CRP > 5, body temperature > 38°C), non-union musculo-tendinous lesion at the time of inclusion.
* Hemophilia, coagulation disorders
* Regular medication intake that may influence the data
* Any metabolic or hormonal disorder. Contraindications to competitive swimming
* Any other condition that the investigating physician considers may pose an individual risk or interfere with the evaluation of the data.

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 58 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in index of coordination (IdC) from motor behavior | each 6 month during 3 years
  To observe the effects of a manipulated swimming frequency or velocity on the coordination (this one was quantified in terms of an index of coordination (IdC) based on the lag time between the propulsive phases of each swimming movement) from motor behavior viewpoints in elite level swimmers and para-swimmers.

SECONDARY OUTCOMES:
Change in energy expenditure by contribution of aerobic and anaerobic metabolism. | each 6 month during 3 years
  To observe the effects of a manipulated swimming frequency or velocity on the variation of in the consumption of oxygen and lactic acid in elite level swimmers and para-swimmers.

CONTACTS AND LOCATIONS:
Overall Officials: Seifert Ludovic, Pr., Principal Investigator — University of Rouen Normandie
Locations (1):
- Institut National du Sport, de l'Expertise et de la Performance, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thompson KG, Haljand R, MacLaren DP. An analysis of selected kinematic variables in national and elite male and female 100-m and 200-m breaststroke swimmers. J Sports Sci. 2000 Jun;18(6):421-31. doi: 10.1080/02640410050074359. PMID 10902677
- [Background] Thompson KG, MacLaren DP, Lees A, Atkinson G. The effects of changing pace on metabolism and stroke characteristics during high-speed breaststroke swimming. J Sports Sci. 2004 Feb;22(2):149-57. doi: 10.1080/02640410310001641467. PMID 14998093
- [Background] Seifert L, Chollet D, Rouard A. Swimming constraints and arm coordination. Hum Mov Sci. 2007 Feb;26(1):68-86. doi: 10.1016/j.humov.2006.09.003. Epub 2006 Nov 28. PMID 17126942
- [Background] Seifert L, Komar J, Crettenand F, Millet G. Coordination pattern adaptability: energy cost of degenerate behaviors. PLoS One. 2014 Sep 25;9(9):e107839. doi: 10.1371/journal.pone.0107839. eCollection 2014. PMID 25255016
- [Background] Seifert L, Komar J, Araujo D, Davids K. Neurobiological degeneracy: A key property for functional adaptations of perception and action to constraints. Neurosci Biobehav Rev. 2016 Oct;69:159-65. doi: 10.1016/j.neubiorev.2016.08.006. Epub 2016 Aug 6. PMID 27506266
- [Background] Ribeiro J, Toubekis AG, Figueiredo P, de Jesus K, Toussaint HM, Alves F, Vilas-Boas JP, Fernandes RJ. Biophysical Determinants of Front-Crawl Swimming at Moderate and Severe Intensities. Int J Sports Physiol Perform. 2017 Feb;12(2):241-246. doi: 10.1123/ijspp.2015-0766. Epub 2016 Aug 24. PMID 27248207
- See also: Description of the project — https://www.univ-rouen.fr/actualites/neptune-un-projet-de-recherche-laureat-de-lappel-a-projets-sport-de-tres-haute-performance/